CLINICAL TRIAL: NCT04669626
Title: The Ability of Octenilin® to Reduce Odour of Malodorous Wound - a Single-center Randomized Double Blinded Controlled Pilot Study
Brief Title: The Ability of Octenilin® to Reduce Odour of Malodorous Wound
Acronym: Odour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Odour
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Wound; Wound Heal
Keywords: Odour; wound care
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 2 (Other): Wound cleansing with NaCl (natrium chlorid) solution 0.9%
  Interventions: Other: Use of NaCl 0.9%
- Group 1 (Experimental): Wound cleansing with Octenilin®
  Interventions: Other: Use of Ocetnilin

INTERVENTIONS:
Other: Use of Ocetnilin — Visits to the outpatient wound-care centre as directed by a physician. Wound care performed by the respective study nurse according to the study-protocol. Each dressing change will be the same and will be as follows:
  * Removal of old dressing
  * Applying a soaked gaze with Octenilin® on the wound (5 minutes)
  * Mechanical debridement if necessary
  * Wound cleansing with Octenilin®
  * Application of new dressing (according to the wound healing phases, medical prescription)
  Arms: Group 1
Other: Use of NaCl 0.9% — Visits to the outpatient wound-care centre as directed by a physician. Wound care performed by the respective study nurse according to the study-protocol. Each dressing change will be the same and will be as follows:
  * Removal of old dressing
  * Applying a soaked gaze with NaCl 0.9% solution on the wound (5 minutes)
  * Mechanical debridement if necessary
  * Wound cleansing with NaCl 0.9% solution
  * Application of new dressing (according to the wound healing phases, medical prescription)
  Arms: Group 2

SUMMARY:
Malodours are a common complication of chronic wounds. They are the result of the proliferation of aerobic and anaerobic micro-organisms on the wound surface, where they metabolize healthy tissue which leads to the production of sloughy and even necrotic tissue. Wound odour has a big impact on the quality of life of patients.

Currently the standard of care for the management of malodourous wounds are systemic antibiotics, absorbent wound dressings with or without activated carbon and, topical antimicrobials. The application of topical antimicrobials such as antiseptics against wound odour is part of the standard care. One suggested antiseptic in a recent published standard is Octenilin®. There is ample anecdotal evidence about the efficacy of Octenilin® in reducing wound odour. Therefore, we propose here to document this ability by evaluating the odour of wounds washed with Octenilin® versus standard care (NaCl 0.9% solution).

DETAILED DESCRIPTION:
Malodours are a common complication of chronic wounds. They are the result of the proliferation of aerobic and anaerobic micro-organisms on the wound surface, where they metabolize healthy tissue which leads to the production of sloughy and even necrotic tissue. Wound odour has a big impact on the quality of life of patients. Patients describe living with a chronic malodourous wound as devastating particularly in respect to social interaction. The key to addressing the negative consequences of malodorous and/or discharging wounds is an effective wound managements plan based on accurate and holistic assessment of the patient and the wound.

Currently the standard of care for the management of malodourous wounds are systemic antibiotics, absorbent wound dressings with or without activated carbon and, topical antimicrobials. The application of topical antimicrobials such as antiseptics against wound odour is part of the standard care. One suggested antiseptic in a recent published standard is Octenilin®. Octenilin® wound cleansing solution is on the Swiss market since 2006 and is routinely used in outpatient wound care centers. It exhibits good performance in the reduction of biofilm's pathogens and has excellent moisturizing properties. While there is ample anecdotal evidence about the efficacy of Octenilin® in reducing wound odour, we propose here to document this ability by evaluating the odour of wounds washed with Octenilin® versus standard care (NaCl 0.9% solution).

ELIGIBILITY:
Inclusion Criteria:

* A chronic malodourous wound
* Age over 18 years
* Proficiency in the French language

Exclusion Criteria:

* Valid informed consent is not or cannot be given
* Patients needing dressings with Silver
* Patients needing charcoal dressings
* Patients under antibiotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Assessment of wound odour | 12 weeks
  assessment of wound odour intensity by the study nurse using a Visual Analog Scale (VAS) from 0 to 100 (perceived odour).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Probst, Prof Dr, Principal Investigator — HES-SO University of Applied Sciences and Arts Western Switzerland
Locations (1):
- Cité Génération Maison de santé, Onex, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
data will be ananymised